CLINICAL TRIAL: NCT01244230
Title: An Open-label, Uncontrolled 4-week Study to Assess the Safety, Efficacy and Pharmacokinetics of Allegra® (Dry Syrup Formulation) 15 mg or 30 mg Twice Daily in Pediatric Patients With Atopic Dermatitis
Brief Title: Safety, Efficacy and Pharmacokinetic Study of Allegra in Pediatric Patients With Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFY10718; U1111-1115-4048 (Other: UTN)
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Age 6 months - 2 years (Experimental): Patients between 6 months and 2 years old - Type: Experimental
  Interventions: Drug: fexofenadine/Allegra (M016455)
- Age 2 - 11 years (Experimental): Patients between 2 and 11 years (and under 10.5 kg)
  Interventions: Drug: fexofenadine/Allegra (M016455)
- Age 2 - 11 years (and over 10.5 kg) (Experimental): Patients between 2 and 11 years (and over 10.5 kg)
  Interventions: Drug: fexofenadine/Allegra (M016455)

INTERVENTIONS:
Drug: fexofenadine/Allegra (M016455) — Pharmaceutical form:dry syrup formulation to be suspended in water
  Route of administration: oral

SUMMARY:
Primary Objective:

To evaluate safety (4 weeks)

Secondary Objectives:

* To evaluate the long-term safety (12 weeks)
* To evaluate the efficacy
* To characterize the pharmacokinetic profile

DETAILED DESCRIPTION:
The study consists of four phases: up to 9-day screening phase, main 4-week treatment phase, up-to 8-week extension phase, and up-to 5-day post-treatment phase.

ELIGIBILITY:
Inclusion criteria:

* Aged 6 months through 11 years
* Patients with atopic dermatitis

Exclusion criteria:

* Main itching scores are 4 or less than 2 on last three consecutive days before registration.
* Patients who have itching only on face, head, or diaper area.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 4 weeks
The number of clinically significant abnormalities for laboratory findings | 4 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events | 12 weeks
The number of clinically significant abnormalities for laboratory findings | 12 weeks
Changes from baseline in main itching scores on patient diary | 4 weeks
Changes from baseline in pruritus intensity scores assessed by investigator or subinvestigator | week 2 and 4
Pharmacokinetic parameters of fexofenadine at steady state; AUC | week 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Japan (13):
  - Investigational Site Number 392012, Hitachi-Naka
  - Investigational Site Number 392001, Isumi
  - Investigational Site Number 392010, Itoshima-Shi
  - Investigational Site Number 392002, Katsushika-ku
  - Investigational Site Number 392006, Kofu
  - Investigational Site Number 392011, Komae-Shi
  - Investigational Site Number 392007, Komatsu-Shi
  - Investigational Site Number 392003, Kōtoku
  - Investigational Site Number 392013, Nagano
  - Investigational Site Number 392009, Okayama
  - Investigational Site Number 392008, Osaka
  - Investigational Site Number 392004, Setagaya-Ku
  - Investigational Site Number 392005, Setagaya-Ku